CLINICAL TRIAL: NCT06725589
Title: Brain Network Connectivity of Patients With Metabolic Diseases
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-706-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertension, T2DM, obesity, gout, and patients without the above diseases: hypertension, T2DM, obesity, gout, and patients without the above diseases
  Interventions: Other: metabolic disease

INTERVENTIONS:
Other: metabolic disease — metabolic disease

SUMMARY:
The global prevalence of metabolic diseases, including hypertension, type 2 T2DM mellitus (T2DM), gout and obesity, has risen over the past two decades. Brain controls human behavior and metabolism in organisms. It will be very interesting to explore whether there are similarities or relations among different metabolic diseases and how brain might be involved in the progression of different metabolic diseases.

We analyzed the PET-CT images and clinical biological markers of 112 cases of hypertension, 56 cases of T2DM, 11 cases of obesity, 14 cases of gout, and 497 cases without the above diseases. Standardized uptake value ratios (SUVRs) were extracted from different brain regions according to AAL brain atlas using Spatial-Normalization-of-Brain-PET-Images. Partial correlation analysis was used to analyze the correlation of the SUVRs of different brain regions with clinical biological markers by controlling sex, age and BMI. Brain network metabolic connectivity was analyzed using Permutation_IHEP software and visualized using BrainNet Viewer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent brain PET-CT in Sun Yat-sen Memorial Hospital from January 2018 to June 2024

Exclusion Criteria:

* Brain lesions, including patients with brain atrophy, cerebral ischemia and trauma, epilepsy, brain tumors, brain trauma, and psychiatric disorders; Patients with missing medical history or brain imaging data; Patients with tumor.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent brain PET-CT examination in Sun Yat-sen Memorial Hospital from January 2018 to June 2024 and met our inclusion and exclusion criteria were included in the analysis. About 690 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
the correlation between metabolic changes in different brain regions and blood test results in patients without metabolic diseases, hypertension, T2DM, gout and obesity | 2024.01-2024.06

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, China